CLINICAL TRIAL: NCT01862874
Title: A Phase III Placebo-controlled Clinical Trial to Study the Tolerability, Immunogenicity and Efficacy of V501 in 16- to 26-year-old Japanese Men
Brief Title: Efficacy and Tolerability Study of V501 in Japanese Males (V501-122)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V501-122; 132237 (Registry Identifier: JAPIC-CTI); 2015-002931-16 (EudraCT Number); V501-122 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Anogenital Human Papilloma Virus Infection; Condyloma Acuminata
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V501 (Experimental): Participants received V501 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Follow-up was up to Month 36.
  Interventions: Biological: V501
- Placebo (Placebo Comparator): Participants received placebo 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Follow-up was up to Month 36.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V501 — Formulated with aluminum hydroxyphosphate sulfate (AAHS) adjuvant
  Other Names: GARDASIL™; Quadrivalent HPV (Type 6, 11, 16 and 18) L1 Virus-Like Particle vaccine
  Arms: V501
Biological: Placebo — Formulated with AAHS adjuvant
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy and tolerability of V501 (quadrivalent Human Papilloma Virus [HPV] [Type 6, 11, 16 and 18] L1 Virus-Like Particle vaccine, GARDASIL™) in healthy, 16- to 26-year old Japanese males. The hypotheses tested are: 1) V501 reduces the combined incidence of HPV 6-, 11-, 16-, or 18-related persistent infection compared with placebo, and 2) V501 reduces the combined incidence of HPV 6-, 11-, 16-, or 18-related persistent infection, condyloma acuminata, penile/perianal/perineal intraepithelial neoplasia, or penile, perianal, or perineal cancer compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Japanese
* No clinical evidence of gross genital lesion suggesting sexually-transmitted disease and no clinically present external genital warts
* Other inclusion criteria will be discussed with the investigator during screening

Exclusion Criteria:

* History of known prior vaccination with an HPV vaccine or plans to receive one outside the study
* History of external genital warts
* History of severe allergic reaction that required medical intervention
* Received immune globulin or blood-derived products in the past 6 months or plan to receive any before Month 7 of the study
* History of splenectomy, is currently immunocompromised, or has been diagnosed with immunodeficiency, Human Immunodeficiency Virus (HIV), lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition
* Received immunosuppressive therapy in the past year, excluding inhaled, nasal, or topical corticosteroids and certain regimens of systemic corticosteroids
* Known thrombocytopenia or coagulation disorder that would contraindicate intramuscular injections
* Ongoing alcohol or drug abuse within the past 12 months

Ages: 16 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1124 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mikamo H, Yamagishi Y, Murata S, Yokokawa R, Han SR, Wakana A, Sawata M, Tanaka Y. Efficacy, safety, and immunogenicity of a quadrivalent HPV vaccine in Japanese men: A randomized, Phase 3, placebo-controlled study. Vaccine. 2019 Mar 14;37(12):1651-1658. doi: 10.1016/j.vaccine.2019.01.069. Epub 2019 Feb 20. PMID 30797638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1129 participants were screened and 1124 were randomized.
Period: Overall Study
Arm/Group | V501 | Placebo
Started | 562 (Randomized participants) | 562 (Randomized participants)
Vaccination 1 | 561 | 562
Vaccination 2 | 539 | 542
Vaccination 3 | 530 | 532
Completed | 483 | 485
Not Completed | 79 | 77
Not completed — Randomized not treated | 1 | 0
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 26 | 29
Not completed — Physician Decision | 5 | 3
Not completed — Withdrawn by parent/guardian | 1 | 1
Not completed — Withdrawal by Subject | 46 | 40
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V501 | Placebo | Total
Number analyzed (Participants) | 562 | 562 | 1124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.6 (2.1) | 22.6 (2.0) | 22.6 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 562 | 562 | 1124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 562 | 562 | 1124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Combined Incidence of HPV Type 6, 11, 16, or 18-related Persistent Infection
Description: Persistent infection was defined as 1) polymerase chain reaction (PCR) positive to HPV Type 6, 11, 16, or 18 in 2 consecutive anogenital or biopsy samples collected ≥4 months apart, or 2) Pathology Panel consensus diagnosis of condyloma acuminate, penile/perianal/perineal intraepithelial neoplasia (PIN), penile, perianal, or perineal cancer and PCR detection of HPV Type 6, 11, 16, or 18 in an adjacent section and PCR positive for the same HPV type at a separate adjacent visit. The combined incidence of HPV Type 6, 11, 16, or 18 persistent infection detected in samples from ≥2 consecutive visits ≥6 months apart was assessed.
Time Frame: Up to Month 36
Population: Participants who were seronegative at Day 1 and PCR negative from Day 1 through Month 7 to the relevant HPV type, received all 3 vaccinations, did not deviate from the study protocol in ways that might interfere with vaccine efficacy, and had ≥1 follow-up visit after Month 7.
Measure: Number; unit: Cases per 100 person-years of follow-up
Units Other Than Participants: Person-years follow-up
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 497 | 498
Number analyzed (Person-years follow-up) | 1137 | 1123
Cases per 100 person-years of follow-up | 0.3 | 1.9
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority; p < 0.001, One-sided exact test; Vaccine Efficacy = 85.9, 95% CI 2-sided [52.7 to 97.3] — Vaccine efficacy is defined as the percentage reduction in relative risk for the V501 group versus the placebo group; If the lower bound of the 95% confidence interval for vaccine efficacy excludes 0%, then superiority of the V501 group is demonstrated

2. Primary Outcome: Percentage of Participants With Maximum Temperature ≥37.5°C Reported on the Vaccination Report Card
Description: Body temperature (oral or oral equivalent) was recorded on the Vaccination Report Card (VRC). The percentage of participants with a maximum temperature ≥37.5°C was summarized.
Time Frame: Up to 5 days after any vaccination
Population: Participants who received ≥1 study vaccination and had follow-up data available.
Measure: Number; unit: Percentage of participants
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 551 | 557
Percentage of participants | 2.7 | 3.9
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Other — Statistical testing of no difference in incidence of maximum temperature ≥37.5°C; p = 0.256, Miettinen & Nurminen; Risk Difference (RD) = -1.2, 95% CI 2-sided [-3.5 to 0.9] — Risk difference (V501 - placebo) was estimated using the Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants With an Injection-site Adverse Event Prompted on the Vaccination Report Card
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study drug. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug or a protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study drug or protocol-specified procedure is also an AE. The percentage of participants with an injection-site AE prompted on the VRC (erythema, pain, and swelling) was summarized.
Time Frame: Up to 5 days after any vaccination
Population: Participants who received ≥1 study vaccination and had follow-up data available.
Measure: Number; unit: Percentage of participants
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 554 | 559
Percentage of participants
  Injection-site erythema | 24.5 | 21.6
  Injection-site pain | 54.9 | 48.5
  Injection-site swelling | 21.3 | 14.5
Statistical Analysis 1: Comparison: V501 vs Placebo; Injection-site erythema; Test type: Other — Statistical testing of no difference in incidence of injection-site erythema; p = 0.251, Miettinen & Nurminen; Risk Difference (RD) = 2.9, 95% CI 2-sided [-2.1 to 7.9] — Risk difference (V501 - placebo) was estimated using the Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V501 vs Placebo; Injection-site pain; Test type: Other — Statistical testing of no difference in incidence of injection-site pain; p = 0.033, Miettinen & Nurminen; Risk Difference (RD) = 6.4, 95% CI 2-sided [0.5 to 12.2] — Risk difference (V501 - placebo) was estimated using the Miettinen & Nurminen method
Statistical Analysis 3: Comparison: V501 vs Placebo; Injection-site swelling; Test type: Other — Statistical testing of no difference in incidence of injection-site swelling; p = 0.003, Miettinen & Nurminen; Risk Difference (RD) = 6.8, 95% CI 2-sided [2.3 to 11.3] — Risk difference (V501 - placebo) was estimated using the Miettinen & Nurminen method

4. Primary Outcome: Percentage of Participants With a Systemic Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study drug. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug or a protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study drug or protocol-specified procedure is also an AE. The percentage of participants with a systemic AE was summarized.
Time Frame: Up to 15 days after any vaccination
Population: Participants who received ≥1 study vaccination and had follow-up data available.
Measure: Number; unit: Percentage of participants
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 554 | 559
Percentage of participants | 14.4 | 15.4
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Other — Statistical testing of no difference in incidence of systemic AEs; Risk Difference (RD) = -0.9, 95% CI 2-sided [-5.2 to 3.3] — Risk difference (V501 - placebo) was estimated using the Miettinen & Nurminen method

5. Primary Outcome: Percentage of Participants With a Vaccine-related Systemic Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study drug. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug or a protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study drug or protocol-specified procedure is also an AE. Vaccine-related AEs are those that were deemed possibly, probably, or definitely related to vaccine administration by the investigator. The percentage of participants with a vaccine-related systemic AE was summarized.
Time Frame: Up to 15 days after any vaccination
Population: Participants who received ≥1 study vaccination and had follow-up data available.
Measure: Number; unit: Percentage of participants
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 554 | 559
Percentage of participants | 3.4 | 5.0
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Other — Statistical testing of no difference in incidence of vaccine-related systemic AEs; Risk Difference (RD) = -1.6, 95% CI 2-sided [-4.1 to 0.8] — Risk difference (V501 - placebo) was estimated using the Miettinen & Nurminen method

6. Secondary Outcome: Combined Incidence of HPV Type 6, 11, 16, or 18-related Persistent Infection or Disease
Description: Persistent infection was defined as 1) polymerase chain reaction (PCR) positive to HPV Type 6, 11, 16, or 18 in 2 consecutive anogenital or biopsy samples collected ≥4 months apart, or 2) Pathology Panel consensus diagnosis of condyloma acuminate, penile/perianal/perineal intraepithelial neoplasia (PIN), penile, perianal, or perineal cancer and PCR detection of HPV Type 6, 11, 16, or 18 in an adjacent section and PCR positive for the same HPV type at a separate adjacent visit. The incidence of persistent infection detected in samples from ≥2 consecutive visits ≥6 months apart was assessed. Disease was defined as HPV Type 6, 11, 16, or 18-related condyloma acuminate, PIN, penile, perianal, or perineal cancer. The combined incidence of HPV Type 6, 11, 16, or 18 persistent infection or disease was assessed.
Time Frame: Up to Month 36
Population: as for outcome 1
Measure: Number; unit: Cases per 100 person-years at risk
Units Other Than Participants: Person-years follow-up
Arm/Group | V501 | Placebo
Number analyzed (Participants) | 498 | 498
Number analyzed (Person-years follow-up) | 1148 | 1132
Cases per 100 person-years at risk | 0.3 | 1.9
Statistical Analysis 1: Comparison: V501 vs Placebo; Test type: Superiority; p < 0.001, One-sided exact test; Vaccine Efficacy = 86.5, 95% CI 2-sided [55.2 to 97.4] — Vaccine efficacy is defined as the percentage reduction in relative risk for the V501 versus the placebo group; If the lower bound of the 95% confidence interval for vaccine efficacy excludes 0%, superiority of the V501 group is demonstrated

ADVERSE EVENTS:
Time Frame: Up to 36 months
Description: The at-risk population was participants who received ≥1 study vaccination and had follow-up data available
Arm/Group | V501 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/554 | 1/559
Serious Adverse Events (participants affected / at risk) | 0/554 | 1/559
Other Adverse Events (participants affected / at risk) | 329/554 | 303/559
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V501 (N=554) | Placebo (N=559)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V501 (N=554) | Placebo (N=559)
Injection-site erythema (General disorders) | 137 (217) | 122 (179)
Injection-site pain (General disorders) | 304 (563) | 271 (480)
Injection-site swelling (General disorders) | 118 (181) | 82 (121)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT01862874/Prot_SAP_000.pdf